CLINICAL TRIAL: NCT01486446
Title: Phase 2a, Exploratory, Double-blind, Placebo-controlled Two-part Study to Evaluate the Safety, Efficacy, Tolerability and Pharmacokinetics of Topically Applied XPF-002 (XEN402 8% w/w Ointment) in Patients With Primary/Inherited Erythromelalgia
Brief Title: Phase 2a, Exploratory Study to Evaluate the Safety, Efficacy, Tolerability and Pharmacokinetics of XPF-002 in Patients With Primary/Inherited Erythromelalgia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XPF-002-202
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Primary Erythromelalgia; Inherited Erythromelalgia
Keywords: IEM; EM; Erythromelalgia; Erythermalgia; Red neuralgia; Peripheral Vascular Disease; Vascular Disease; Cardiovascular Disease
MeSH Terms: conditions — Erythromelalgia; Peripheral Vascular Diseases; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XPF-002 (Experimental): XEN402 8% w/w ointment for topical application, applied to the skin twice daily for 14 or 21 days
  Interventions: Drug: XPF-002
- Placebo (Placebo Comparator): XEN402 0% w/w ointment for topical application. Identical content and appearance to the XPF-002 ointment but without the active medicine. Applied to the skin twice daily for 14 or 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XPF-002 — XEN402 8% w/w ointment for topical application, applied to the skin twice daily for 14 or 21 days
  Arms: XPF-002
Drug: Placebo — XEN402 0% w/w ointment for topical application. Identical content and appearance to the XPF-002 ointment but without the active medicine. Applied to the skin twice daily for 14 or 21 days.
  Arms: Placebo

SUMMARY:
This is a Phase 2a single-center, randomized, double-blind, Placebo-controlled, parallel group study with XPF-002 applied twice daily over 14 or 21 days in patients with Primary/Inherited Erythromelalgia (IEM). The purpose of this study is to determine whether XPF-002 is safe and effective in the treatment of pain caused by IEM.

DETAILED DESCRIPTION:
Your role in the study would include:

* Travelling to the clinic (in Anniston, Alabama, USA) for 3 out-patient visits, each lasting approximately 1 day
* Travelling and staying in the clinic for 2 in-patient stays:
* For the first in-patient visit you will have to spend 8 days and 7 nights in the clinic
* For the second in-patient visit you will have to spend 2 days and 1 night in the clinic You can bring books, laptops and DVDs to the clinic.

If you do not live within driving distance to the clinic you will need to stay in the local area (in Anniston, at a local hotel) for 1 to 2 weeks while you use the ointment, in addition to the in-patient portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have a Body Mass Index (BMI) of 18-40 kg/m2 (inclusive)
* Have primary or inherited erythromelalgia (IEM)
* Experience flares of pain in your feet or hands caused by erythromelalgia
* Be generally healthy (apart from your pain)
* Stop taking your usual pain medications and certain other medications for up to 11.5 weeks
* Not be pregnant or breast-feeding
* Must be able and willing to provide informed consent and willing to comply with all study procedures and restrictions

Exclusion Criteria:

* Must not be in constant pain (must not continually be in moderate pain, 3/10 or more)
* Coexistent source of pain from other conditions that may interfere with the study interpretation
* HIV, Hepatitis B or C
* Treatment for significant depression within 6 months of Screening
* Not willing to use adequate contraception
* Alcoholism, alcohol or substance abuse
* Presence or history of major psychiatric disturbance
* Any other condition or finding that may pose undue risk for participation
* Use of any other investigational drug in the 30 days prior to dosing
* Donation or loss of whole blood or plasma prior to dosing as follows: 50 mL to 499 mL within 30 days, or more than 499 mL within 56 days
* Employee or relative of an employee who is directly involved in the study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Almena L Free, MD, Principal Investigator — Pinnacle Research Group LLC.
Locations (1):
- Pinnacle Research Group, LLC., Anniston, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | XPF-002 | Placebo
Started | 7 | 1
Completed | 6 | 1
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XPF-002 | Placebo | Total
Number analyzed (Participants) | 7 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 0 | 6
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (19.3) | 77 (NA) — Only 1 placebo subject, therefore no SD. | 44.4 (22.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 1 | 8

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Average Cooling Duration (Minutes Per Day) for EM-related Pain in Treatment Period 2
Description: Using diary cards, subjects recorded the use and duration of all non-pharmacological cooling methods used to relieve their EM pain each day during Treatment Period 2.
  A smaller average duration of cooling each day in Treatment Period 2 indicates that subjects were in less pain/required less use of cooling to relieve their EM pain and vice versa.
Time Frame: 14-21 Days
Measure: Mean (Inter-Quartile Range); unit: minutes/day
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 7 | 1
minutes/day | 7.8 [0 to 13.3] | 86 [NA to NA] — Only 1 placebo subject, therefore no IQR.

2. Other Pre Specified Outcome: Time to Exit (Minutes) From Standard Heat Inductions in Treatment Period 1, Compared to Baseline
Description: A standard heat induction was performed on multiple occasions pre-and post treatment. Subjects placed their feet in front of an electric heater for up to 75 minutes. Subjects rated their pain intensity/severity using numerical and categorical rating scales at fixed intervals before, during and after the heating procedure.
  The heating procedure continued until one of the pre-defined stopping criteria were met, or when the 75 minutes were over. Subjects could stop the procedure at any time if pain was intolerable. A stopwatch was used to record the time the heating procedure was stopped. This time is known as "Time to Exit".
  A longer Time to Exit compared to Baseline indicates that subjects were able to tolerate the heat for a longer period when on treatment.
Time Frame: Baseline to Day 5
Measure: Mean (Inter-Quartile Range); unit: Percentage of Baseline
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 7 | 1
Percentage of Baseline | 138 [78 to 188] | 96 [NA to NA] — Only 1 placebo subject, therefore no IQR.

3. Primary Outcome: Average Daily Use of Cooling for Erythromelalgia-Related Pain in Treatment Period 2
Description: Using diary cards, subjects recorded the use of all non-pharmacological cooling methods used to relieve their erythromelalgia (EM) pain each day during Treatment Period 2.
  A smaller average number of cooling uses each day in Treatment Period 2 indicates that subjects were in less pain/required less use of cooling to relieve their EM pain and vice versa.
Time Frame: 14-21 Days
Measure: Mean (Inter-Quartile Range); unit: cooling uses/day
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 7 | 1
cooling uses/day | 0.24 [0.03 to 0.27] | 2.4 [NA to NA] — Only 1 placebo subject, therefore no IQR.

4. Other Pre Specified Outcome: Time to Exit (Minutes) From Standard Heat Inductions in Treatment Period 2, Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and 14 or 21 days
Measure: Mean (Inter-Quartile Range); unit: Percentage of Baseline
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 7 | 1
Percentage of Baseline | 100 [92 to 112] | 107 [NA to NA] — Only 1 placebo subject, therefore no IQR.

5. Other Pre Specified Outcome: Time to Moderate Pain (Minutes) During Standard Heat Inductions in Treatment Period 1, Compared to Baseline
Description: A standard heat induction was performed on multiple occasions pre-and post treatment. Subjects placed their feet in front of an electric heater for up to 75 minutes. Subjects rated their pain intensity/severity using numerical and categorical rating scales at fixed intervals before, during and after the heating procedure.
  The heating procedure continued until one of the pre-defined stopping criteria were met, or when the 75 minutes were over. Subjects could stop the procedure at any time if pain was intolerable.
  A stopwatch was used to record the time the subject recorded a pain intensity numerical score of 5 or more (on a scale of 0-10). This time is known as "Time to Moderate Pain".
  A longer Time to Moderate Pain compared to Baseline indicates that subjects were able to tolerate the heat for a longer period when on treatment.
Time Frame: Baseline to Day 5
Measure: Mean (Inter-Quartile Range); unit: Percentage of Baseline
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 7 | 1
Percentage of Baseline | 137 [74 to 172] | 90 [NA to NA] — Only 1 placebo subject, therefore no IQR.

6. Other Pre Specified Outcome: Time to Moderate Pain (Minutes) During Standard Heat Inductions in Treatment Period 2, Compared to Baseline
Description: as for outcome 5
Time Frame: Baseline and 14 or 21 days
Measure: Mean (Inter-Quartile Range); unit: Percentage of Baseline
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 7 | 1
Percentage of Baseline | 103 [91 to 115] | 135 [NA to NA] — Only 1 placebo subject, therefore no IQR.

7. Other Pre Specified Outcome: Daily Pain (Maximum Pain Intensity) in Treatment Period 2, Compared to Baseline
Description: During Baseline and Treatment Period 2, subjects recorded pain scores in their diary cards 3 times each day (upon waking, lunchtime and evening).
  On each recording occasion, subjects recorded the maximum pain experienced since the previous recording occasion using an 11 point numerical rating scale of pain intensity, PINRS (where 0 = no pain and 10 = worst pain imaginable).
  A lower score compared to Baseline indicates that the subjects experienced less severe pain on treatment than during Baseline.
Time Frame: Baseline to 14 or 21 days
Measure: Mean (Inter-Quartile Range); unit: Percentage of Baseline
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 7 | 1
Percentage of Baseline | 78.5 [75.9 to 94.2] | 76 [NA to NA] — Only 1 placebo subject, therefore there is no IQR.

8. Other Pre Specified Outcome: Sleep Interference Due to Pain in Treatment Period 2, Compared to Baseline
Description: During Baseline and Treatment Period 2, subjects recorded sleep interference scores in their diary cards for each night (scores were recorded upon waking).
  Sleep Interference due to pain is scored using an 11 point numerical rating scale where 0 = pain does not interfere with sleep and 10 = completely interferes, unable to sleep due to pain.
  A lower sleep interference score compared to Baseline indicates that the subjects' pain interfered with sleep less on treatment than during Baseline.
Time Frame: Baseline to 14 or 21 days
Measure: Mean (Inter-Quartile Range); unit: Percentage of Baseline
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 7 | 1
Percentage of Baseline | 76.5 [48.8 to 86.9] | 46 [NA to NA] — Only 1 placebo subject, therefore no IQR.

ADVERSE EVENTS:
Arm/Group | XPF-002 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/1
Other Adverse Events (participants affected / at risk) | 7/7 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XPF-002 (N=7) | Placebo (N=1)
Hospitalization due to worsening erythromelalgia pain (Vascular disorders) | 1 (1) | 0 (0) — Subject was admitted to hospital for treatment of worsening erythromelalgia pain 131 days following their last dose of study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XPF-002 (N=7) | Placebo (N=1)
Headache (Nervous system disorders) | 3 (8) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (3) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Nodule (General disorders) | 1 (4) | 0 (0)
Flushing (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oopharyngeal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Tooth infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (3) | 0 (0)
Cyanosis (Vascular disorders) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This was a small trial with many exploratory efficacy measures. There was no primary outcome measure, all measures are "other: pre-specified".

Only 8 subjects were enrolled (1 placebo), the actual number of Adverse Events is used, not incidence.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days